CLINICAL TRIAL: NCT04694781
Title: An Open Label, Phase 1 Trial of LVGN6051 as Single Agent and in Combination With Pembrolizumab in Advanced or Metastatic Malignancy
Brief Title: Study of LVGN6051 (CD137 Agonist Antibody) in Advanced or Metastatic Malignancy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lyvgen Biopharma Holdings Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LVGN6051-201
Record Dates: First submitted 2020-12-16; First posted 2021-01-05 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-03

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Monotherapy Dose Escalation (Experimental): LVGN6051 monotherapy dose escalation
  Interventions: Drug: LVGN6051
- Monotherapy Dose Expansion (Experimental): LVGN6051 dose expansion cohorts
  Interventions: Drug: LVGN6051
- Combination therapy dose escalation (Experimental): LVGN6051 in combination with anti-PD-1 antibody pembrolizumab dose escalation
  Interventions: Drug: LVGN6051; Drug: Pembrolizumab
- Combination therapy dose expansion (Experimental): LVGN6051 in combination with anti-PD-1 antibody pembrolizumab dose expansion cohorts
  Interventions: Drug: LVGN6051; Drug: Pembrolizumab

INTERVENTIONS:
Drug: LVGN6051 — Route of administration is IV infusion, and the frequency of administration is once every 3 weeks (Q3W). one cycle is 3 weeks, and treatment can be up to 35 cycles if patients receive benefits.
Drug: Pembrolizumab — Route of administration is IV infusion, and the frequency of administration is once every 3 weeks (Q3W). one cycle is 3 weeks, and treatment can be up to 35 cycles if patients receive benefits.
  Arms: Combination therapy dose escalation; Combination therapy dose expansion

SUMMARY:
The study of LVGN6051-201 is designed to use a bridging dose escalation to quickly establish the maximum tolerated dose (MTD) and/or the recommended dose for expansion (RDE) as well as the recommended Phase 2 dose(s) (RP2D) of LVGN6051, both as a single agent (monotherapy) and in combination with a fixed dose of anti-PD-1 antibody (Pembrolizumab) in the treatment of advanced or metastatic malignancy.

DETAILED DESCRIPTION:
Based on the dose escalation results from the study of LVGN6051-101, a bridging dose escalation (3+3) is used in study of LVGN6051-201. The traditional 3 + 3 dose escalation algorithm to identify the MTD and/or RDE and RP2D of LVGN6051 as a single agent (monotherapy) and in combination with pembrolizumab. The first stage of the study is the single agent dose escalation and expansion phase (Part A). The second stage of the study is the combination dose escalation and expansion phase (Part B). Patients will be considered evaluable for safety and tolerability if they receive at least one dose of LVGN6051 or pembrolizumab at the specified cohort dose. Patients in all parts of the trial will remain on therapy until confirmed disease progression or for 2 years, whichever occurs first. However, patients who are clinically unstable will discontinue following the initial assessment of disease progression

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged ≥ 18 years.
* Ability to understand and willingness to sign a written informed consent document.
* Patients must have a histologically or cytologically confirmed metastatic or unresectable malignancy.
* Estimated life expectancy, in the judgment of the Investigator, of at least 90 days.
* Adequate bone marrow, liver, and renal functions.
* Men and women of childbearing potential must agree to take highly effective contraceptive methods.
* Patients should recover from all reversible AEs of previous anticancer therapies to baseline.

Exclusion Criteria:

* Receipt of CD137 and or PD-1 antibodies.
* Receipt of systemic anticancer therapy within 5 half-lives of the first dose of study treatment.
* Known active CNS metastasis and/or carcinomatous meningitis.
* Has received a live-virus vaccine within 30 days.
* Has had a Grade ≥ 3 allergic reaction to treatment with a monoclonal antibody.
* Abnormality of QT interval or syndrome.
* Patients with history of Grade ≥ 3 immune-related AEs (irAEs) or irAE.
* Patients who are receiving an immunologically-based treatment for any reason.
* Active or chronic autoimmune disease that has required systemic treatment in the past 2 years or who are receiving systemic therapy for an autoimmune or inflammatory disease.
* Has a clinically significant cardiac condition, including unstable angina, acute myocardial infarction within 6 months.
* Has an active infection requiring intravenous (i.v.) anti-infectives within 14 days before the first dose of study treatment.
* Tested positive of HIV or HBV or HCV.
* Female patients who are pregnant or breastfeeding.
* Any evidence of severe or uncontrolled systemic disease.
* Has previously had a CAR-T therapy, or stem cell or bone marrow or solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent adverse events (TEAEs) including determination of DLTs and serious AEs (SAEs) | up to 24 months
  Adverse events will be assessed, and severity will be assigned by using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0.
MTD or RDE or RP2D | up to 24 months
  maximal tolerated dose, recommended dose for expansion or recommended phase 2 dose

SECONDARY OUTCOMES:
DCR | up to 24 months
  DCR will be documented as the proportion of patients with best overall response of CR, PR, or stable disease (SD). DCR per RECIST v1.1, iRECIST, and Cheson/Lugano criteria.
PK parameter AUC | up to 24 months
  Area under the serum concentration versus time curve (AUC) will be determined.
PK parameter Cmax | up to 24 months
  Peak Plasma Concentration (Cmax) will be summarized.
PK parameter t1/2 | up to 24 months
  Serum concentration half-life t1/2 will be summarized.
ADA to LVGN6051 | up to 24 months
  The presence of ADA directed against LVGN6051 will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Luo, Study Director — Lyvgen Biopharma
Locations (2):
- China (2):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - Shanghai Chest Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided